CLINICAL TRIAL: NCT03158792
Title: Evaluation of Non-Surgical Venous Thromboembolism Prophylaxis Dosing Strategies: Enoxaparin 20mg Versus 30mg Subcutaneously Once Daily in Elderly Patients With Impaired Renal Function
Brief Title: Enoxaparin 20mg Versus 30mg Subcutaneously Once Daily in Elderly Patients With Impaired Renal Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lebanese American University (Other)
Responsible Party: Principal Investigator, Nibal Chamoun, Clinical Assistant Professor of Pharmacy Practice and Clinical Coordinator, Lebanese American University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LAU.SOP.NC1.25/Jun/2015
Record Dates: First submitted 2017-04-09; First posted 2017-05-18 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Venous Thromboembolism; Renal Impairment
Keywords: Anticoagulation; Thromboprophylaxis; Anti-Xa levels; Elderly; Prevention; Enoxaparin; Low molecular weight heparin
MeSH Terms: conditions — Venous Thromboembolism; Renal Insufficiency | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enoxaparin 20 mg (Active Comparator)
  Interventions: Drug: Enoxaparin 20Mg/0.2mL Prefilled Syringe
- Enoxaparin 30 mg (Active Comparator)
  Interventions: Drug: Enoxaparin 60Mg/0.6Ml Inj Syringe 0.6Ml

INTERVENTIONS:
Drug: Enoxaparin 20Mg/0.2mL Prefilled Syringe — Enoxaparin 20mg subcutaneously once daily
  Arms: Enoxaparin 20 mg
Drug: Enoxaparin 60Mg/0.6Ml Inj Syringe 0.6Ml — Enoxaparin 30mg subcutaneously once daily. Half of the graduated 60Mg/0.6Ml Inj Syringe is administered
  Arms: Enoxaparin 30 mg

SUMMARY:
This is a clinical trial including non-surgical patients, 70 years of age or older, with renal impairment requiring pharmacological venous thromboembolism prevention during hospitalization. Patients are randomized to receive either 20 mg or 30mg of enoxaparin. Both dosing regimens of enoxaparin have been approved for thromboprophylaxis in impaired kidney function in different countries. Therefore, this study aims to evaluate the efficacy and safety of enoxaparin 20mg versus 30mg subcutaneously daily by comparing anti-xa levels, thrombosis and bleeding events.

ELIGIBILITY:
Inclusion Criteria:

* Non-surgical patients
* 70 years of age or older
* With renal impairment (creatinine clearance ≤35ml/min)
* Requiring pharmacological thromboprophylaxis

Exclusion Criteria:

* Indication for a treatment dose of anticoagulant treatment
* Knee surgery or hip surgery within 10 to 35 days, respectively
* Surgery, trauma, hemodialysis, peritoneal dialysis, or bleeding
* History of heparin-induced thrombocytopenia
* Known or suspected hypersensitivity to any component of study drug
* Patients with an excessive risk of bleeding and not eligible for pharmacological thromboprophylaxis based on physician assessment or due to any of the 3 major risk factors including active gastroduodenal ulcer, bleeding within the past three months prior to hospital admission, or a platelet count of <50,000 platelets/ mm3

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-10-24 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Peak anti-Xa levels | Day 3 of thromboprophylaxis
  Peak anti-Xa levels, drawn 4 hours after the enoxaparin dose is given

SECONDARY OUTCOMES:
Trough anti-xa levels | Day 3 of thromboprophylaxis
  Trough anti-Xa levels, drawn right before the third enoxaparin dose is given
Bleeding according to the GUSTO bleeding criteria. | Bleeding within 30 days will be assessed from randomization till date of bleeding or date of discharge, whichever comes first.
Objectively confirmed symptomatic or asymptomatic venous thromboembolism (VTE) including both deep vein thrombosis (DVT) and or pulmonary embolism (PE). | Venous thromboembolism (VTE) within 30 days will be assessed from randomization till date of VTE or date of discharge, whichever comes first.
  Chart documentation of objectively detected DVT by either bilateral venography or duplex ultrasonography whereas PE detection by contrast enhanced computerized tomography scan (CT Scan) or Magnetic resonance imaging (MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Nibal R Chamoun, PharmD, Principal Investigator — Lebanese American University
Locations (1):
- LAU Medical Center-Rizk Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chamoun N, Ghanem H, Hachem A, Hariri E, Lteif C, Mansour H, Dimassi H, Zalloum R, Ghanem G. Evaluation of prophylactic dosages of Enoxaparin in non-surgical elderly patients with renal impairment. BMC Pharmacol Toxicol. 2019 May 7;20(1):27. doi: 10.1186/s40360-019-0308-8. PMID 31064405